CLINICAL TRIAL: NCT01281033
Title: CompariSon of Manual Aspiration With Rheolytic Thrombectomy in Patients Undergoing Primary PCI. The SMART-PCI Trial
Acronym: SMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Careggi Hospital (Other)
Collaborators: Cardiovascular Research Foundation, New York (Other)
Responsible Party: Principal Investigator, David Antoniucci, MD, Careggi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART-PCI
Record Dates: First submitted 2011-01-18; First posted 2011-01-21 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: ST-segment Elevation Myocardial Infarction; Thrombus
Keywords: primary PCI; ST-segment elevation myocardial infarction; thrombus aspiration
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Thrombosis | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- thrombus-aspiration group (Active Comparator): In patients in the thrombus-aspiration group, the thrombus-aspiration is manually performed.
  Interventions: Procedure: Manual Thrombectomy
- AngioJet Rheolytic Thrombectomy (Experimental): AngioJet Rheolytic Thrombectomy (RT) System consists of a drive unit console, disposable pump set, and disposable catheter.
  Interventions: Procedure: AngioJet Rheolytic Thrombectomy (RT) System

INTERVENTIONS:
Procedure: Manual Thrombectomy — In patients in the thrombus-aspiration group, this step is followed by the advancing of the 6-French Export Aspiration Catheter (Medtronic; crossing profile, 0.068 in.) into the target coronary segment during continuous aspiration.
  Other Names: manual aspiration
  Arms: thrombus-aspiration group
Procedure: AngioJet Rheolytic Thrombectomy (RT) System — The AngioJet Rheolytic Thrombectomy (RT) System consists of a drive unit console, disposable pump set, and disposable catheter. Thrombectomy is accomplished by the introduction of a pressurized high velocity saline stream through directed orifices in the catheter distal tip so that thrombus is entrained (Bernoulli effect), dissociated into small particles, and evacuated from the body through the catheter and associated tubing. The pump set consists of a high pressure pulsatile pump which is used to generate the flow necessary for the dissociation and evacuation of thrombus, an effluent bag for the collection and storage of thrombus debris, and associated tubing.
  Other Names: Mechanical Thrombectomy
  Arms: AngioJet Rheolytic Thrombectomy

SUMMARY:
To compare rheolytic thrombectomy (RT) with manual thrombus aspiration (MTA) in patients with acute ST-segment elevation myocardial infarction (STEMI) undergoing primary PCI.

Occlusive thrombosis triggered by a disrupted or eroded atherosclerotic plaque is the anatomic substrate of ST-segment elevation myocardial infarction (STEMI). Due to this substrate, macro- and microembolization during percutaneous coronary intervention (PCI) in AMI is frequent and may result in obstruction of the microvessel network, and decreased efficacy of reperfusion and myocardial salvage. Direct stenting without predilation or postdilation is the most simplistic approach to the problem of embolization, and may decrease embolization and the incidence of the no-reflow phenomenon. Other approaches to the problem of microvessel embolization include thrombectomy before stent implantation, and the use of antiembolic devices (filters and occlusive devices with retrieval of thromboembolic material after stent implantation). Most concluded studies on removing of thrombus before stenting used manual aspiration catheters and meta-analyses derived from these studies support the use of manual thrombus aspiration (MTA) catheters in the setting of primary PCI. MTA is currently recommended in the setting of primary PCI as a Class II b recommendation; level of evidence B. Rheolytic thrombectomy (RT) using multiple jets of saline solution and aspiration based on the Bernoulli effect has been proven to be effective in decreasing major adverse events during PCI in saphenous vein grafts or native coronary arteries with angiographic evidence of thrombus, and 2 out of 3 concluded studies have shown a better reperfusion and clinical outcome in patients randomized to RT as compared to control.

DETAILED DESCRIPTION:
The SMART Study is an on-label, randomized, 2-arms, prospective study in patients with STEMI undergoing primary PCI. Diagnosis of STEMI is based on ECG evidence of ischemic ST changes, clinical symptoms, and elevated CK and CK-MB cardiac enzymes. Patients who are eligible for the Study and who provide written informed consent will be included in the study.

Inclusion Criteria:

* Patient is > 18 years of age.
* Patient has ST-segment elevation of at least 0.1 mV in 2 or more contiguous leads or presumably new LBBB for all types of infarcts.
* Patient's AMI presentation is greater than 30 minutes but less than 6 hours after symptom onset.
* Patient provides written informed consent.
* Patient has no childbearing potential or is not pregnant.
* Target artery has a reference vessel diameter of at least 2.5 mm on visual assessment at baseline angiography.

Exclusion Criteria:

* Known prior history of renal insufficiency (serum creatinine 2.0 mg/dL).
* Cardiogenic shock.
* Prior administration of thrombolysis for the current infarction.
* Participation in another study.
* Major surgery within past 6 weeks.
* History of stroke within 30 days, or any history of hemorrhagic stroke.
* Severe hypertension (systolic BP > 200 mm Hg or diastolic BP > 110 mm Hg) not controlled on antihypertensive therapy.
* Known neutropenia ( <1000 neutrophils per mm3) or known severe thrombocytopenia (< 50,000 platelets per mm3).
* Patient unwilling to receive blood products.
* Previously stented IRA (stent thrombosis).
* Inability to identify the IRA.
* Severe vessel tortuosity that enables OCT assessment.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria:

* Patient is > 18 years of age.
* Patient has ST-segment elevation of at least 0.1 mV in 2 or more contiguous leads or presumably new LBBB for all types of infarcts.
* Patient's AMI presentation is greater than 30 minutes but less than 6 hours after symptom onset.
* Patient provides written informed consent. Patient has no childbearing potential or is not pregnant

Angiographic inclusion criteria:

* All patients with or without evidence of thrombus are eligible.
* Target artery has a reference vessel diameter 2.5 mm on visual assessment at baseline angiography.

Exclusion Criteria:

Clinical exclusion criteria:

* Known prior history of renal insufficiency (serum creatinine 2.0 mg/dL).
* Cardiogenic shock.
* Prior administration of thrombolysis for the current infarction.
* Participation in another study.
* Major surgery within past 6 weeks.
* History of stroke within 30 days, or any history of hemorrhagic stroke.
* Severe hypertension (systolic BP > 200 mm Hg or diastolic BP > 110 mm Hg) not controlled on antihypertensive therapy.
* Known neutropenia ( <1000 neutrophils per mm3) or known severe thrombocytopenia (< 50,000 platelets per mm3).
* Patient unwilling to receive blood products

Angiographic exclusion criteria:

* Previously stented IRA (stent thrombosis).
* Inability to identify the IRA.
* Severe vessel tortuosity that enables OCT assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Post-thrombectomy thrombus burden as assessed by coronary OCT | baseline
  OCT images analysis. The primary end-point of the study will be the number of thrombus containing vascular quadrants considering vascular slices.

SECONDARY OUTCOMES:
Angiographic thrombus grade after thrombectomy | baseline
ST-segment resolution at 30 minutes post-PCI, assessed by 12-lead ECG | 30 minutes
Angiographic markers of reperfusion:TIMI flow grade, TIMI myocardial blush. | baseline
Procedural angiographic complications : distal embolization, no-reflow, perforation, dissection. | baseline
Infarct size and microvascular obstruction measured by MRI at 3-7 days | 3-7 days
Six-month MACE (death, reinfarction, TVR, stroke) | six months
Six-month binary angiographic restenosis (> 50%) | six months
Percent of malapposed struts at 6-month OCT follow-up | six months
Six-month left ventricular remodelling by 2D ECHO | six months
Twelve-month MACE or hospital admission for heart failure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Antoniucci, MD, Principal Investigator — Careggi Hospital, Division of Invasive Cardiology
Locations (1):
- Careggi Hospital, Florence, Italy

REFERENCES:
- [Derived] Parodi G, Valenti R, Migliorini A, Maehara A, Vergara R, Carrabba N, Mintz GS, Antoniucci D. Comparison of manual thrombus aspiration with rheolytic thrombectomy in acute myocardial infarction. Circ Cardiovasc Interv. 2013 Jun;6(3):224-30. doi: 10.1161/CIRCINTERVENTIONS.112.000172. Epub 2013 Jun 4. PMID 23735474